CLINICAL TRIAL: NCT05738460
Title: The Effects of Intrapartum Antibiotic Prophylaxis to Prevent Group B Streptococcal Early-onset Disease on Intestinal Microbiome and Immunity of Offspring
Brief Title: Effects of IAP-EOGBSD on Offspring's Gut Microbiome and Immunity.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zhujiang Hospital (Other)
Collaborators: Zhongshan Bo Ai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMOH2102
Record Dates: First submitted 2023-01-18; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-02

CONDITIONS: Healthy; Metabolism; Microbiome
Keywords: Microbiome,; maternal and offspring; healthy
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reproductive tract GBS colonization group of mothers during pregnancy: Reproductive tract GBS colonization group of mothers during pregnancy，Use of antibiotics
  Interventions: Drug: antibiotics
- No reproductive tract GBS colonization group in mothers during pregnancy: No reproductive tract GBS colonization group in mothers during pregnancy

INTERVENTIONS:
Drug: antibiotics — Reproductive tract GBS colonization group of mothers during pregnancy，Use of antibiotics
  Other Names: antibiotic
  Groups: Reproductive tract GBS colonization group of mothers during pregnancy

SUMMARY:
This study is planned to be recruited in two hospitals in South China, Zhujiang Hospital of Southern Medical University and Zhongshan Boai Hospital Recruit participants, plan to recruit obstetrics and child health departments in study hospitals, meet inclusion and discharge criteria 1~3 infants, a total of 360, recruited by Pearl River Hospital of Southern Medical University and Zhongshan Boai Hospital 180 people each.

DETAILED DESCRIPTION:
This is a case-control study. By collecting fecal samples of infants and young children in the observation group and control group at different time points (0~1 years old, 1~2 years old, 2~3 years old), the intestinal flora of infants and young children was detected by 16S rDNA sequencing, and fecal calprotectin (CP) and secretory IgA (SIgA) were detected by ELISA. To study the effects of exposure factors on intestinal flora and immunity in offspring.

ELIGIBILITY:
Inclusion Criteria:

* Infants:37-41 weeks of age, born through vaginal delivery, 2500g<= birth weight < 4000g,0-3 years of age;
* The mother: birth ranging in age from 18 to 40 years old, the single pregnancy, pregnancy 35 -41 weeks to complete the GBS screening;
* The guardian agrees to participate in the study voluntarily.

Exclusion Criteria:

* Infants and children with serious congenital abnormalities, infections or clinical diseases;
* Antibiotics should be used in infants within 2 weeks, probiotics, prebiotics and biostime should be supplemented, or long-term drug treatment should be given for digestive, immune, blood and other diseases;
* Infant mothers: childbirth after long-term drug treatment due to digestive, immune, blood and chronic diseases during pregnancy; Or infants who were breastfed within 12 hours of antibiotic use after delivery;
* Any medical or non-medical condition that the investigator deems inappropriate to participate in.

Ages: 37 Weeks to 41 Weeks | Sex: All
Age Groups: Child
Study Population: Infants: 37-41 weeks of age, born through vaginal delivery, 2500g<= birth weight < 4000g, 0-3 years of age; 2. The mother: birth ranging in age from 18 to 40 years old, the single pregnancy, pregnancy 35 - 41 weeks to complete the GBS screening; 3. The guardian agrees to participate in the study voluntarily.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Intestinal flora | Fecal samples of infants and young children in the observation group and control group at different time points (0~1 years old) of offspring were collected
  Analyze the effect of intrapartum antibiotics on the prevention of early-onset group B streptococcal diseases on the gut microbiome.
Secretory IgA | Fecal samples of infants and young children in the observation group and control group at different time points (0~1 years old) of offspring were collected
  Analyze the effect of intrapartum antibiotics on the prevention of early-onset group B streptococcal diseases on the secretory IgA of offspring.
Calprotectin | Fecal samples of infants and young children in the observation group and control group at different time points (0~1 years old) of offspring were collected
  Analyze the effect of intrapartum antibiotics on the prevention of early-onset group B streptococcal diseases on the cailprotectin of offspring.

SECONDARY OUTCOMES:
Intestinal flora | Fecal samples of infants and young children in the observation group and control group at different time points 1~2 years of offspring were collected
  Analyze the effect of intrapartum antibiotics on the prevention of early-onset group B streptococcal diseases on the gut microbiome.
Secretory IgA | Fecal samples of infants and young children in the observation group and control group at different time points 1~2 years of offspring were collected
  Analyze the effect of intrapartum antibiotics on the prevention of early-onset group B streptococcal diseases on the secretory IgA of offspring.
Calprotectin | Fecal samples of infants and young children in the observation group and control group at different time points 1~2 years of offspring were collected
  Analyze the effect of intrapartum antibiotics on the prevention of early-onset group B streptococcal diseases on the cailprotectin of offspring.

OTHER OUTCOMES:
Intestinal flora | Fecal samples of infants and young children in the observation group and control group at different time points 2~3 years old of offspring were collected
  Analyze the effect of intrapartum antibiotics on the prevention of early-onset group B streptococcal diseases on the gut microbiome.
Secretory IgA | Fecal samples of infants and young children in the observation group and control group at different time points 2~3 years old of offspring were collected
  Analyze the effect of intrapartum antibiotics on the prevention of early-onset group B streptococcal diseases on the secretory IgA of offspring.
Calprotectin | Fecal samples of infants and young children in the observation group and control group at different time points 2~3 years old of offspring were collected
  Analyze the effect of intrapartum antibiotics on the prevention of early-onset group B streptococcal diseases on the secretory IgA of offspring.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Wang, Study Chair — Southern Medical University, China
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China